CLINICAL TRIAL: NCT01165333
Title: Cilengitide (EMD121974) in Combination With Irradiation in Children and Young Adults With Newly Diagnosed Diffuse Intrinsic Pontine Glioma: Phase I Study
Brief Title: Cilengitide in Combination With Irradiation in Children With Diffuse Intrinsic Pontine Glioma
Acronym: CILENT-0902
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CILENT-0902
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma
Keywords: Paediatric oncology; Cilengitide; Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Cilengitide; Pharmacogenomic Variants; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose escalation (Experimental): In the first part of the trial, a dose-ranging study in ca. 18-21 patients will be done. A standard dose escalation strategy will be used including 3 to 6 patients at each dose level, the first cohort of patients being treated at dose level one Interventions : Cilengitide dose escalation ; Concomitant radiotherapy ; Pharmacokinetic ; Pharmacogenetic
  Interventions: Drug: Cilengitide dose escalation; Radiation: Concomitant radiotherapy; Biological: Pharmacokinetic; Biological: Pharmacogenetic
- Cohort extension (Experimental): An additional 20 patients will be treated at the recommended dose in order to confirm the recommended cilengitide dose and to carry out the exploratory investigations Interventions : Cilengitide ; Concomitant radiotherapy ; Pharmacokinetic ; Pharmacogenetic
  Interventions: Drug: Cilengitide; Radiation: Concomitant radiotherapy; Biological: Pharmacokinetic; Biological: Pharmacogenetic; Biological: Exploratory investigation

INTERVENTIONS:
Drug: Cilengitide dose escalation — Cilengitide will be administered intravenously over 60 minutes, twice a week, at a given dose.
  The Cilengitide dose (mg/m²/infusion)levels are as follows :
  * 240
  * 480
  * 720
  * 1200
  * 1800
  Other Names: Cilengitidine
  Arms: Dose escalation
Drug: Cilengitide — Patients will be treated at the recommended dose in order to confirm the recommended cilengitide dose and to carry out the exploratory investigations
  Other Names: cilengitidine
  Arms: Cohort extension
Radiation: Concomitant radiotherapy — 1.8 Gy per fraction for a total of 54 Gy over 6 weeks, from monday to friday of the first cycle. The radiation will imperatively begin between 3 and 7hours after the end of Cilengitide infusion.
Biological: Pharmacokinetic — A pharmacokinetic assessment for Cilengitide will be carried for all patients. The pharmacokinetic (PK) samples will be drawn during day 1 and day 2 of the first cycle of treatment.
Biological: Pharmacogenetic — For every patient 1 blood sample will be taken before study treatment. These blood samples can be made at any hour of the day, and does not require to be taken on an empty stomach. DNA will be extracted in the Laboratory of Pharmacology.Constitutional polymorphisms of genes will be measured before the treatment initiation.
Biological: Exploratory investigation — Evaluate the metabolic impact of the treatment with dynamic MRI (diffusion, perfusion, spectro), and with FDG-PETand sestamibi SPECT.
  Arms: Cohort extension

SUMMARY:
The aim of the study is to determine the safety of Cilengitide in combination with radiation therapy.

DETAILED DESCRIPTION:
The prognosis of children and young adults with a malignant glioma in the brain stem or a recurrent malignant glioma (in whatever site) is very poor. Over the last few decades, many therapeutic trials have been performed but have failed to significantly improve survival in these patients. There is thus a need to test new drugs in these indications. There is a strong biological rationale for the use of anti-angiogenic drugs in high-grade glioma. Cilengitide (EMD121974; Merck KgaA, Darmstadt, Germany), a cyclic pentapeptide containing the sequence RGD (cyclo-[Arg-Gly-Asp-Dphe-(NmeVal)]) is a selective antagonist of integrins αvβ3 and αvβ5, which are strongly involved in tumour angiogenesis. Positive results with Cilengitide in preclinical models of glioblastoma, its particularly attractive safety profile and its encouraging efficacy in phase I and II studies in adults and children make it a potentially effective molecule for the treatment of malignant glioma in children. Furthermore, its combination with radiotherapy to be appears synergistic, without any apparent increase in toxicity.

In this study, Cilengitide will be evaluated when concurrently administered with radiotherapy as a first-line treatment and then as a maintenance monotherapy in children and young adults with malignant brain stem glioma. The main objective will be to determine the maximum tolerated dose (MTD) of Cilengitide when administered twice weekly as a 60-minute intra-venous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diffuse intrinsic pontine glioma
* Metastatic disease allowed
* MRI measurable disease according to the WHO criteria and for extension cohort

  * Patient is able to undergo functional MRI (diffusion, perfusion, spectro)
  * Patient is able to undergo FDG-PET and sestamibi SPECT
* Life expectancy > 8 weeks after the start of study treatment.
* No prior chemotherapy for the present cancer; no treatment for any other cancer during the last 5 years.
* No prior cerebral radiation therapy
* Age > 6 months and < 21 years
* Lansky Play Scale > 50 or ECOG Performance Status < 2; NB: Children and young adults with a worse performance status due to glioma-related motor paresis can be included.
* Absolute neutrophils count > 1.5 x 109/l, Platelets > 100 x 109/l
* Total bilirubin < 1,5 x ULN, AST and ALT< 2,5 x ULN
* Serum creatinine ≤ 1,5 X ULN for age. If serum creatinine > 1,5 ULN, creatinine clearance must be > 70 ml/min/1.73 m² (EDTA radioisotope GFR or 24 hours urines collection)
* Normal coagulation tests : prothrombin rate (prothrombin time = PT), TCA (PTT), fibrinogen
* No current organ toxicity > grade 2 according to the NCICTCAE version 4.0, especially cardiovascular or renal disease (nephrotic syndrome, glomerulopathy, uncontrolled high blood pressure despite adequate treatment). In case of known or possible cardiac disease, a cardiological advice will be required prior to the inclusion in the study
* If anticonvulsants are currently administered, the dosing regimen must be stable within 1 week prior to the first dose of Cilengitide
* If corticosteroids are administered, the dosing regimen must be stable ≥ 5 days prior to the first dose of Cilengitide.
* Effective contraception for patients (male and female) of reproductive potential during their entire participation in the study and during 6 months after the last administration of Cilengitide.
* Negative pregnancy test (serum beta-HCG) within 1 week prior to start of study treatment in females of reproductive potential
* Patient covered by government health insurance
* Written informed consent given by patient and/or parents/ guardians prior to the study participation

Exclusion Criteria:

* Inclusion criteria failure
* History of coagulation disorder associated with bleeding or recurrent thrombotic events.
* Prior anti-angiogenic therapy
* Any other concomitant anti-cancer treatment not foreseen by this protocol.
* Concomitant inclusion in another therapeutic clinical trial; participation in another therapeutic clinical trial during the last 30 days.
* Pregnancy or breast feeding woman
* Uncontrolled intercurrent illness or active infection
* Unable for medical follow-up (geographic, social or mental reasons)

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Determination of the Maximal Tolerated Dose of Cilengitide | After 6 weeks of treatment
  A DLT is defined below:
  Hematological toxicity:
  * grade 4 neutropenia for more than 5 days
  * grade 3 or 4 neutropenia with documented infection
  * grade 3 or 4 thrombopenia for more than 5 days
  * requirement of platelet transfusion support for more than 5 days
  Non-hematological toxicity:
  Any grade 3 or 4 non-hematological toxicity of whatever duration with the exception of (i) nausea/vomiting without appropriate treatment, and (ii)isolated, transient fever occurring outside an episode of neutropenia), with the exclusion of toxicities related to any other well-identified cause.

SECONDARY OUTCOMES:
Safety profile of the Cilengitide | During all the study
  toxicities (NCI-CTCAE v4.0)
study of the pharmacoKinetic profile of Cilengitide | Day 1 and 2 of first cycle
  Blood samples of 2 mL will be collected at each time point : before Cilengitide infusion, at the end of infusion, 30 mn after the end of infusion, 60 mn, 90 mn, 2 hrs, 4 hrs, 6 hrs, 24 hrs after the end of infusion
estimate efficacy in terms of response according to histopathology | Every 3 cycles
  WHO criteria
Progression-free and overall survival | During all the study
  6-month-PFS overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LEBLOND, MD, Principal Investigator — Centre Oscar Lambret
Locations (9):
- France (9):
  - Hôpital des Enfants, Groupe Hospitalier, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU, Hôpital d'Enfants de la Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Institut Curie, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU, Toulouse
  - Institut Gustave-Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No